CLINICAL TRIAL: NCT01176591
Title: Human Behavioral Pharmacology Laboratory (HBPL) Study of the Impact of the NK1 Antagonist Aprepitant (Emend®) on Stress-Induced Cocaine and Alcohol Craving
Brief Title: HBPL Study of the Impact of the NK1 Antagonist Aprepitant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 811184; K01DA025073 (NIH)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Cocaine Dependence; Alcohol Dependence
Keywords: Cocaine and alcohol dependence (CAD)
MeSH Terms: conditions — Cocaine-Related Disorders; Alcoholism | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Session 1, Aprepitant Session 2 (Experimental): Participants receive placebo in session 1 and Aprepitant in session 2 of a psychological stressor presentation and receive placebo in session 1 and Aprepitant in session 2 of a physiological stressor presentation. Participants take Aprepitant (80 mg) or placebo tablets for 7 days prior to each session.
  Interventions: Drug: Placebo session 1, Aprepitant session 2
- Placebo Session 1, Placebo Session 2 (Placebo Comparator): Participants receive placebo in session 1 and placebo in session 2 of a psychological stressor presentation and receive placebo in session 1 and placebo in session 2 of a physiological stressor presentation. Participants take placebo tablets for 7 days prior to each session. The placebo group is used for analysis purposes in order to control for any order effects found in the Experimental group.
  Interventions: Drug: Placebo session 1, Placebo session 2

INTERVENTIONS:
Drug: Placebo session 1, Aprepitant session 2 — placebo in session 1, Aprepitant 80 mg in session 2, oral administration.
  Other Names: Aprepitant
  Arms: Placebo Session 1, Aprepitant Session 2
Drug: Placebo session 1, Placebo session 2 — Placebo, one per session, oral administration
  Other Names: Placebo
  Arms: Placebo Session 1, Placebo Session 2

SUMMARY:
The proposed research will focus on investigating the determinants and consequences of CAD via measurement of physiological, behavioral and subjective effects of physiologic and psychologic stress cues in CAD volunteers in the laboratory, and through examination of the effects of the effects of Aprepitant, an NK1 antagonist, on the above effects. This study will examine the effects of the above stress cues on cocaine and alcohol craving under acute Aprepitant dosing, and under placebo conditions. The study is a within-subjects crossover design using 24 subjects.

DETAILED DESCRIPTION:
Non treatment seeking subjects with DSM IV cocaine and alcohol dependence were included. Subjects received double-blind acute dosing of 80 mg of aprepitant (Emend) at session start, or matched placebo. During each session subjects were exposed to one of two types of stressors, one stressor per session, presented in counterbalanced order across participants. The Physiologic stress was the cold-pressor task. Subjects immersed their hand in cold water for up to 3 minutes. The psychological stress was the Trier Social Stress Test it was completed in 25 minutes: 5 min audio taped instructions, 10 min to mentally prepare for their performance tasks, 5 min to complete a public speaking task and 5 min to complete a mental arithmetic task. Outcome measures included: Alcohol Craving measured by visual analog scale, cocaine craving measured by visual analog scale and The Multiple Choice Procedure. Each assessment was done during study screening, and then at multiple times during each study session.

ELIGIBILITY:
Inclusion Criteria

1. Male or female and 18 years of age to 60
2. The subject has used cocaine and alcohol at least once per month for at least the past year, and has used cocaine and alcohol within 30 days prior to signing consent.
3. Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
4. Understands and signs the informed consent.

Exclusion Criteria:

1. Meets Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria for current dependence on any substance other than nicotine, cocaine ,alcohol or marijuana
2. Subjects who test positive on the urine drug screen for any illicit drugs other than cocaine and marijuana during screening will be allowed a single retest. Those individuals who test positive for amphetamine during screening, given that they provide a copy of a prescription, will only be included if they can safely discontinue amphetamine use for the duration of the study. Subjects will need to provide a urine free of all illicit drugs other than cocaine and marijuana at study onset to be randomized. Subjects who test positive for any drugs other than marijuana prior to a study session will be allowed a single retest and a chance to reschedule their session. If the subject tests positive for any drug other than marijuana at the retest, their participation in the study will be terminated.
3. Subjects who meet current or lifetime DSM-IV criteria for bipolar affective disorder, schizophrenia, or any psychotic disorder
4. Current severe psychiatric symptoms- (e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring anti-depressant therapy) as diagnosed using the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID), the Hamilton Anxiety Rating Scale (Ham A), and Hamilton Rating Scale for Depression (HAM-D).
5. Individuals scoring > 10 on the Hamilton Rating Scale for Depression (HAM-D).
6. Use of any investigational medication within the past 30 days.
7. Concomitant treatment with psychotropic medications or prescription opioids.
8. Concomitant use of any one of the following drugs or classes of drugs:

   Reserpine Verapamil theophylline, trimethoprim, cimetidine, haloperidol, benzodiazepines, or antiepileptic drugs (AEDs).
9. Patients with a known hypersensitivity to aprepitant.
10. Patients with severe concurrent illnesses such as bronchospastic disease, hyperthyroidism, diabetes mellitus.
11. Patients with known AIDS or other serious illnesses that may require hospitalization during the study.
12. Female subjects who are pregnant or lactating, or female subjects of child-bearing potential who are not using acceptable methods of birth control; acceptable methods of birth control include:

    Barrier method (diaphragm or condom) with spermicide Intrauterine progesterone contraceptive system Levonorgestrel implant Medroxyprogesterone acetate contraceptive injection, or Oral contraceptives.
13. Patients with impaired renal function, as indicated by corrected creatinine clearance below 60 ml/min as determined by the modified Cockcroft equation (CDC, 1986).
14. An unacceptable liver panel or liver function tests (LFTs) that may be indicative of hepatic dysfunction.
15. Clinical laboratory tests (e.g., complete blood count (CBC), blood chemistries, urinalysis) outside normal limits, as determined by the study PI.
16. History of significant heart disease or dysfunction (e.g., an arrhythmia which required medication, Wolff Parkinson -White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure).
17. Electrocardiography (EKG) indicative of 1st degree heart block, sinus tachycardia, left-axis deviation, non-specific ST or T-wave changes.
18. History of chest pain associated with cocaine use that prompted a visit to a physician.
19. Any medical or psychological condition that could jeopardize the subject's safe participation in the trial as determined by the PI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, MD, Study Director — Perelman School of Medicine
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Session 1, Aprepitant Session 2: Placebo in session 1; Aprepitant: 80 mg in session 2, oral administration.
- Placebo in Session 1, Placebo in Session 2: Placebo, one per session, oral administration
Period: Session 1
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo in Session 1, Placebo in Session 2
Started | 10 | 3
Completed | 10 | 3
Not Completed | 0 | 0
Period: Session 2
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo in Session 1, Placebo in Session 2
Started | 10 | 3
Completed | 10 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Session1, Placebo Session 2: Placebo, one per session, oral administration
- Total: Total of all reporting groups
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session1, Placebo Session 2 | Total
Number analyzed (Participants) | 10 | 3 | 13
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 3 | 13
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Craving as Measured on the Visual Analog Scale (VAS) 1
Description: The VAS is a 100 mm line anchored at both ends. Participants mark where on the line their craving falls, with closer to 0 indicating less craving, and closer to 100 indicating more craving. Data are analyzed by using a ruler to determine the actual mm value of the participant mark.
Time Frame: Session 1
Population: Comparing Placebo to Placebo
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo Session 1, Placebo Session 2: Placebo in Session 1, Placebo in Session 2, oral administration
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
units on a scale | 19 [0 to 95] | 48 [1 to 100]
Statistical Analysis 1: Comparison: Placebo Session 1, Aprepitant Session 2 vs Placebo Session 1, Placebo Session 2; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

2. Primary Outcome: Alcohol Craving as Measured by the Visual Analog Scale (VAS) 1
Description: as for outcome 1
Time Frame: Session 1
Population: Comparing Placebo to Placebo
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo Session 1, Aprepitant Session 2: Placebo session 1, Aprepitant 80 mg session 2, oral administration.
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
units on a scale | 26.25 [0 to 94] | 38.92 [2 to 100]
Statistical Analysis 1: Comparison: Placebo Session 1, Aprepitant Session 2 vs Placebo Session 1, Placebo Session 2; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

3. Primary Outcome: Cocaine Craving as Measured on the Visual Analog Scale (VAS) 2
Description: as for outcome 1
Time Frame: Session 2
Population: Comparing Aprepitant to Placebo
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
units on a scale | 20 [0 to 84] | 4 [0 to 10]
Statistical Analysis 1: Comparison: Placebo Session 1, Aprepitant Session 2 vs Placebo Session 1, Placebo Session 2; Test type: Superiority or Other; p = 0.046, t-test, 2 sided

4. Primary Outcome: Alcohol Craving as Measured by the Visual Analog Scale (VAS) 2
Description: as for outcome 1
Time Frame: Session 2
Population: Comparing Aprepitant to Placebo
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
units on a scale | 33.22 [0 to 84] | 0.17 [0 to 0.5]
Statistical Analysis 1: Comparison: Placebo Session 1, Aprepitant Session 2 vs Placebo Session 1, Placebo Session 2; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

5. Secondary Outcome: Multiple Choice Procedure (MCP) 1
Description: The MCP measures the relative reinforcing value of a hypothetical single dose of cocaine, as compared to various monetary values. The lower the monetary value where participants switch from preferring cocaine to preferring money, the less value they place on cocaine. MCP findings of cocaine devaluation typically correlate with cocaine abstinence in clinical trials.
Time Frame: Session 1
Population: Comparing Placebo to Placebo
Measure: Mean (Full Range); unit: dollars
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
dollars | 8.58 [0.75 to 20] | 17.33 [12 to 20]

6. Secondary Outcome: Multiple Choice Procedure (MCP) 2
Description: as for outcome 5
Time Frame: Session 2
Population: Comparing Aprepitant to Placebo
Measure: Mean (Full Range); unit: dollars
Arm/Group | Placebo Session 1, Aprepitant Session 2 | Placebo Session 1, Placebo Session 2
Number analyzed (Participants) | 10 | 3
dollars | 7.59 [0.75 to 16] | 17.33 [12 to 20]
Statistical Analysis 1: Comparison: Placebo Session 1, Aprepitant Session 2 vs Placebo Session 1, Placebo Session 2; Test type: Superiority or Other; p = 0.035, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Participants reported adverse events to nurse at each study visit, based on a list of known adverse events and novel adverse events were also recorded.
Groups:
- Placebo Session1, Aprepitant Session 2: Placebo in session 1; Aprepitant: 80 mg in session 2, oral administration
Arm/Group | Placebo Session1, Aprepitant Session 2 | Placebo Session1, Placebo Session 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No